CLINICAL TRIAL: NCT00019682
Title: A Phase III Multi-Institutional Randomized Study of Immunization With the gp100: 209-217 (210M) Peptide Followed by High Dose IL-2 vs. High Dose IL-2 Alone in Patients With Metastatic Melanoma
Brief Title: Aldesleukin With or Without Vaccine Therapy in Treating Patients With Locally Advanced or Metastatic Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2012-02897; NCI-2012-02897 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000066963; 99-C-0051 (Other: IU Health Goshen Center for Cancer Care); T98-0085 (Other: CTEP); NCT00001801 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Recurrent Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; gp100 Melanoma Antigen; montanide ISA 51

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (aldesleukin) (Experimental): Patients receive aldesleukin IV over 15 minutes every 8 hours for 12 doses. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease 3 weeks after completing 2 courses may receive a maximum of 12 additional courses. Patients with complete response may receive a maximum of 2 additional courses.
  Interventions: Biological: Aldesleukin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis
- Arm II (gp100 antigen in Montanide IDA-51 and aldesleukin) (Experimental): Patients receive gp100 antigen emulsified in Montanide ISA-51 SC on day 1. Patients also receive aldesleukin as in Arm I beginning on day 2. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease 3 weeks after completing 2 courses may receive a maximum of 12 additional courses. Patients with complete response may receive a maximum of 2 additional courses.
  Interventions: Biological: Aldesleukin; Biological: gp100 Antigen; Drug: Montanide ISA 51 VG; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: Ro-236019
Biological: gp100 Antigen — Given SC
  Other Names: gp 100; gp100
  Arms: Arm II (gp100 antigen in Montanide IDA-51 and aldesleukin)
Drug: Montanide ISA 51 VG — Given SC
  Arms: Arm II (gp100 antigen in Montanide IDA-51 and aldesleukin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase III trial studies aldesleukin with vaccine therapy to see how well it works compared to aldesleukin alone in treating patients with melanoma that has spread from where it started to nearby tissue or lymph nodes or to other places in the body. Aldesleukin may stimulate a person's white blood cells to kill melanoma cells. Vaccines may make the body build an immune response to kill tumor cells. It is not yet known whether combining aldesleukin with vaccine therapy is more effective than aldesleukin alone in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify whether the addition of the peptide vaccine to high dose interleukin (IL)-2 (aldesleukin) can result in a clinical response rate which may be superior to that found in similar patients treated with high dose IL-2 alone.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile of patients treated on this trial, according to the regimen received.

II. To compare the disease free/progression free survival of patients treated on both arms of the study.

III. To determine the immunologic response experienced by patients who have received the peptide vaccination, as measured by changes in T-cell precursors from before to after treatment.

IV. To evaluate the quality of life of patients before and after high-dose IL-2.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive aldesleukin intravenously (IV) over 15 minutes every 8 hours for 12 doses.

ARM II: Patients receive gp100 antigen emulsified in Montanide ISA-51 subcutaneously (SC) on day 1. Patients also receive aldesleukin as in Arm I beginning on day 2.

In both arms, treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease 3 weeks after completing 2 courses may receive a maximum of 12 additional courses. Patients with complete response may receive a maximum of 2 additional courses.

After completion of treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with measurable metastatic (stage IV or locally advanced stage III) cutaneous melanoma and an expected survival of greater than three months will be considered
* Serum creatinine of 1.6 mg/dl or less
* Total bilirubin 1.6 mg/dl or less
* White blood cell (WBC) 3000/mm^3 or greater
* Platelet count 90,000 mm^3 or greater
* Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less then three times normal
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients of both genders must be willing to practice effective birth control during this trial
* Pathologic confirmation of cutaneous melanoma; patients may enter the study with a pathologic diagnosis of cutaneous melanoma from any institution; all slides will be reviewed at National Institutes of Health (NIH) (department of Anatomic Pathology) and if the diagnosis is not confirmed, the patient will be excluded from the study
* Tissue type human leukocyte antigen (HLA) A0201

Exclusion Criteria:

* Patients who have types of melanoma other than cutaneous, i.e. ocular or mucosal
* Patients who are undergoing or have undergone in the past 4 weeks any other form of therapy except surgery for their cancer, including radiation therapy to any site
* Patients who have active systemic infections, coagulation disorders, autoimmune disease or history of other major medical illnesses such as insulin dependent diabetes mellitus, cardiac ischemia, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary diseases and inflammatory bowel disorders
* Patients who have significant psychiatric disease which in the opinion of the principal investigator would prevent adequate informed consent or render immunotherapy unsafe or contraindicated
* Patients who require steroid therapy or steroid-containing compounds, or have used systemic steroids in the past 4 weeks, or have used topical or inhalational steroids in the past 2 weeks
* Patients who are pregnant
* Patients who are known to be positive for viral hepatitis B or C (hepatitis B surface antigen [HBsAg] or anti hepatitis C virus [HCV]) or human immunodeficiency virus (HIV) (HIV antibody)
* Patients who have any form of primary or secondary immunodeficiency
* Patients who have received previous high dose IL-2 (> 600,000 IU/kg)
* Patients who have received previous gp100 vaccines
* Patients who have an abnormal stress cardiac test (stress thallium, stress multi gated acquisition scan [MUGA], dobutamine echocardiogram or other stress test that will rule out cardiac ischemia)
* Patients who have abnormal pulmonary function tests (forced expiratory volume in one second [FEV1] < 65% or forced vital capacity [FVC] < 65% of predicted)
* Patients who have brain metastasis or history of brain metastasis
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 1999-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Schwartzentruber, Principal Investigator — IU Health Goshen Center for Cancer Care
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Kaiser Permanente Medical Center, Riverside, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - IU Health Goshen Center for Cancer Care, Goshen, Indiana
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - National Institutes of Health, Bethesda, Maryland
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Schwartzentruber DJ, Lawson DH, Richards JM, Conry RM, Miller DM, Treisman J, Gailani F, Riley L, Conlon K, Pockaj B, Kendra KL, White RL, Gonzalez R, Kuzel TM, Curti B, Leming PD, Whitman ED, Balkissoon J, Reintgen DS, Kaufman H, Marincola FM, Merino MJ, Rosenberg SA, Choyke P, Vena D, Hwu P. gp100 peptide vaccine and interleukin-2 in patients with advanced melanoma. N Engl J Med. 2011 Jun 2;364(22):2119-27. doi: 10.1056/NEJMoa1012863. PMID 21631324

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Aldesleukin) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin)
Started | 94 | 91
Completed | 93 | 85
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Aldesleukin) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin) | Total
Number analyzed (Participants) | 94 | 91 | 185
Age, Continuous [Mean (Full Range); unit: years] | 50.3 [18 to 65] | 46.9 [18 to 65] | 48.6 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 63 | 57 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 93 | 91 | 184
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Response Rate (Partial Response [PR] + Complete Response [CR])
Description: A complete response (CR) was defined as the disappearance of all clinical evidence of disease for at least 4 weeks. A partial response (PR) was defined as a 50% or greater decrease in the sum of the products of perpendicular diameters of all measurable lesions for at least one month. No new lesions could appear, and none could increase 25% or more.
Time Frame: Up to 12 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Aldesleukin) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin)
Number analyzed (Participants) | 93 | 85
Participants | 6 | 14
Statistical Analysis 1: Comparison: Arm I (Aldesleukin) vs Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin); Test type: Superiority; p = 0.035, Chi-squared

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival was compared between groups by means of Kaplan-Meier curves using the log-rank test to evaluate the significance of the difference between the arms.
Time Frame: From the date of randomization until documentation of progression or last follow up, assessed up to 12 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Aldesleukin) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin)
Number analyzed (Participants) | 94 | 91
months | 1.6 [1.5 to 1.8] | 2.2 [1.7 to 3.9]
Statistical Analysis 1: Comparison: Arm I (Aldesleukin) vs Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin); Test type: Superiority; p = 0.008, Log Rank — Unadjusted 2 tail p value

3. Secondary Outcome: Change in T-cell Precursors
Description: To measure change in T-cell precursors, PBMC were tested for reactivity by measuring gamma-interferon release after overnight coculture with peptide pulsed T2 cells. PBMC obtained after 4 cycles of study treatment were compared to pre treatment PBMC. A positive assay was defined as greater than 100pg/ml gamma-interferon release and at least twice the release (including all control peptides) by post treatment PBMC compared to pre treatment PBMC.
Time Frame: Baseline to up to 12 years
Population: All patients with paired cryopreserved peripheral blood lymphocytes obtained before any treatment and after completing 4 cycles of treatment.
Measure: Number; unit: Participants with a positive assay
Arm/Group | Arm I (Aldesleukin) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin)
Number analyzed (Participants) | 12 | 37
Participants with a positive assay | 0 | 7
Statistical Analysis 1: Comparison: Arm I (Aldesleukin) vs Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin); Test type: Superiority; p > 0.05, Fisher Exact

4. Secondary Outcome: Change in Quality of Life (QOL) Score Assessed by the FACT-G (Functional Assessment of Cancer Therapy- General), FACT-F (Functional Assessment of Cancer Therapy- Fatigue), SF-36 (Short Form 36) and SDS (Symptom Distress Scale)
Description: QOL was measured before and after 2 cycles of treatment using 4 measures: FACT-G is a 27 item measure of QOL. A total score is calculated by summing across responses on a 5 point scale and ranges from 0-135, with higher scores indicating better QOL. FACT-F is 13 item measure of fatigue. A total score is calculated by summing across responses on a 5 point scale. Total score ranges from 0-52, with higher scores indicating less fatigue. SF-36 is a 36 item measure of self-reported health status. SF-36 is comprised of 8 subscales: physical function, role physical, bodily pain vitality, role emotional function, mental health, social function and general health. Summated scores range from 0-100, with higher scores indicating a better health state. SDS is a 13 item measure of symptom distress. A total score is calculated by summing across responses on a 5 point scale. Total score ranges from 13 to 65, with higher scores indicating more symptom distress.
Time Frame: Baseline to up to 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Aldesleukin) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin)
Number analyzed (Participants) | 93 | 85
units on a scale
  Pre treatment FACT-G | 84.2 (2.77) | 83.8 (2.74)
  Post treatment FACT-G | 76.4 (2.75) | 81.2 (2.71)
  Pre treatment FACT-F | 43.1 (1.47) | 41.5 (1.42)
  Post treatment FACT-F | 36.1 (1.78) | 36.3 (1.73)
  Pre treatment SF-36 | 49.1 (1.93) | 46.6 (1.85)
  Post treatment SF-36 | 42.6 (1.94) | 42.9 (1.89)
  Pre treatment SDS | 21.3 (1.05) | 21.2 (1.05)
  Post treatment SDS | 24.6 (1.17) | 22.8 (1.17)
Statistical Analysis 1: Comparison: Arm I (Aldesleukin) vs Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin); FACT-G scale; Test type: Non-Inferiority — Evaluated inferiority in quality of life outcomes between arms; p > 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Arm I (Aldesleukin) vs Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin); FACT-F scale; Test type: Non-Inferiority — Evaluated inferiority in quality of life outcomes between arms; p > 0.05, Mixed Models Analysis
Statistical Analysis 3: Comparison: Arm I (Aldesleukin) vs Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin); SF-36 scale; Test type: Non-Inferiority — Evaluated inferiority in quality of life outcomes between arms; p > 0.05, Mixed Models Analysis
Statistical Analysis 4: Comparison: Arm I (Aldesleukin) vs Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin); SDS scale; Test type: Non-Inferiority — Evaluated inferiority in quality of life outcomes between arms; p > 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Description: NCI Common Toxicity Criteria Version 2.0 were used for adverse event monitoring. For reporting purposes the individual toxicities were grouped under their respective headings.
Arm/Group | Arm I (Aldesleukin) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin)
Serious Adverse Events (participants affected / at risk) | 1/93 | 2/85
Other Adverse Events (participants affected / at risk) | 93/93 | 85/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Aldesleukin) (N=93) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin) (N=85)
Death (General disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Aldesleukin) (N=93) | Arm II (gp100 Antigen in Montanide IDA-51 and Aldesleukin) (N=85)
Blood or bone marrow (Blood and lymphatic system disorders) | 33 | 41
Arrhythmia (Cardiac disorders) | 4 | 16
General (Cardiac disorders) | 25 | 31
Constitutional symptoms (General disorders) | 15 | 24
Skin (Skin and subcutaneous tissue disorders) | 6 | 6
Gastrointestinal (Gastrointestinal disorders) | 17 | 18
Hepatic (Hepatobiliary disorders) | 36 | 34
Infection or febrile neutropenia (Infections and infestations) | 6 | 7
Metabolic or laboratory-testing result (Metabolism and nutrition disorders) | 19 | 36
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 | 6
Neurologic (Nervous system disorders) | 11 | 22
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 19 | 19
Pain (General disorders) | 10 | 11
Renal or genitourinary (Renal and urinary disorders) | 14 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less